CLINICAL TRIAL: NCT04660565
Title: Belimumab Treatment for IgG4-related Disease, a Prospective, Open-label Clinical Trial
Brief Title: Belimumab Treatment for IgG4-related Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgG4-related disease,Belimumab
Record Dates: First submitted 2020-09-23; First posted 2020-12-09 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Prednisone; belimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid monotherapy Group (Experimental): Patients treated with single glucocorticoid
  Interventions: Drug: Prednisone
- Combination therapy Group (Experimental): Patients treated with Belimumab and glucocorticoid
  Interventions: Drug: Prednisone and Belimumab

INTERVENTIONS:
Drug: Prednisone and Belimumab — Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks to equal to or less than 5mg per day in 3 months. Belimumab will start at the same time as the prednisone induction.
  Other Names: Belimumab treatment
  Arms: Combination therapy Group
Drug: Prednisone — Prednisone/prednisolone: started at 0.6-0. 8mg/kg.d for 2 to 4 weeks, tapered at 5mg per 1-2 weeks to equal to or less than 5mg per day in 3 months.
  Other Names: Prednisone Monotherapy
  Arms: Glucocorticoid monotherapy Group

SUMMARY:
Even though glucocorticoid is the current first line medication for IgG4-RD, it is well accepted in the field that excessive dosage of GC, especially accumulative dosage, is associated with increasing organ damage. Although B cell depletion with rituximab has been verified to be an effective treatment for IgG4-RD, even without concomitant GC therapy, rituximab can increase the risk of infection during the treatment. Belimumab is an IgG1-lambda monoclonal antibody that prevents the survival of B lymphocytes by blocking the binding of soluble human B lymphocyte stimulator protein (BLyS) to receptors on B lymphocytes. Previous studies and trails suggested that the activity of B-cell mediated immunity and autoimmune responses were ameliorated after belimumab without increasing rates of adverse events when compared to standard of care . However, the efficacy and tolerability of belimumab in IgG4-RD patients have not been examined before. This randomized, control clinical trial aimed to evaluate the tolerability and the efficacy of Belimumab for maintenance treatment for IgG4-RD.

DETAILED DESCRIPTION:
IgG4-RD is associated with substantial morbidity and mortality, but there is no established therapy other than GCs for an acute flare. Up to date, no randomized prospective controlled studies have been performed for this disease, and no approved therapy is available. Although GCs are widely and effectively used for treatment of initial disease and flare, they are associated with substantial toxicity which limits their long-term use. Disease flares also occur in many patients either during the GC taper or after GC discontinuation. Patients need a treatment that will more effectively control their disease and avoid GC toxicity. This study will establish the safety and tolerability of Belimumab in IgG4-RD and its ability to reduce the risk of disease flares. There are currently no medicinal products approved for the treatment of IgG4-RD. The majority of cases follow a relapsing course that can lead to permanent tissue damage with attendant morbidity and potential mortality. Glucocorticoids are widely and effectively used for treatment of initial disease and of flare, but they do not prevent recurrence of active disease after their discontinuation and are associated with substantial toxicity. Patients also continue to relapse on the off-label steroid-sparing immunosuppressive medications used by some physicians to manage patients with IgG4-RD; thus, there is a high unmet medical need for more effective therapies in this patient population.

The pathogenesis of IgG4-RD suggests that B-cell depletion may be an effective avenue for therapeutic intervention. Therapeutic depletion of B cells with rituximab reduces disease-relevant biomarkers and appears to have clinical benefit in uncontrolled, retrospective and prospective clinical studies. This study aims to define the efficacy and safety of Belimumab for the prevention of flares of this rare disease. In addition, the potential of Belimumab for minimizing GC exposure could limit the well-known adverse effects of GCs on bone, skin, muscle, adrenal gland, and eyes, and GC association with weight gain, diabetes, hypertension, and neuropsychiatric effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, ≥ 18 years of age at time of informed consent.
2. Written informed consent.
3. Fulfillment of the 2019 ACR/EULAR classification criteria, involving at least one of the following organs: pancreas, lacrimal glands, salivary glands, bile ducts/biliary, orbits, lungs, retroperitoneum, aorta, kidneys, or thyroid gland.
4. New onset or experiencing an IgG4-RD flare that requires initiation or continuation of GC treatment at the time of informed consent. This GC therapy can either be newly initiated or be increased from a maintenance dose of ≤ 10 mg/day of prednisone or equivalent.

Exclusion Criteria:

1. Severe organ dysfunction.
2. Severe infection.
3. Having known immunodeficiency disorder.
4. History of malignancy within the last 10 years.
5. Receipt of any biologic therapy, including B cell-depleting therapy (eg, rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab) or other biologic immunomodulatory agent (abatacept) in the 6 months prior to screening.
6. Non-biologic DMARDs or immunosuppressive agent other than GCs (eg, Leflunomide, Cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, others) have been used withing 12 weeks before screening.
7. Being pregnant, lactating, or planning to become pregnant within 6 months of the test.
8. Positive test for hepatitis B or HIV infection. Positive test for hepatitis B include detection of hepatitis B surface antigen (HBsAg) or HBV-DNA.
9. Chest image ,PPD or TB-ELISPOT results show active tuberculosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Belimumab in reducing the risk of flare in patients with IgG4-RD. | Twelve months
  Relapse was defined as the new progress or recurrence of clinical symptoms or imaging findings with or without IgG4 level re-elevation. the new progress or recurrence of imaging findings were evaluated by MRI, CT or Ultrasound. Primary endpoint is the difference of disease relapse rate between two groups.
The difference of time to first flare between two groups; | Twelve months
  The date of disease flare is defined as the date of initiation of any flare treatment. The date of disease flare is defined as the date of initiation of any flare treatment (new or increased GC treatment, other immunotherapy, or interventional procedure) deemed necessary by the Investigator for the flare.

SECONDARY OUTCOMES:
The effect of Belimumab on disease activity in IgG4-RD patients. | Twelve months
  The estimated treatment effect (ie, the rate ratio of Belimumab versus control), including complete response rate, partial response rate, corresponding 95% CI, and two-sided p-value for the rate ratio will be presented.
Safety and tolerability of Belimumab in patients with IgG4-RD. | Twelve months
  Side effects of Belimumab in patients with IgG4-RD will be evaluated, such as infection, hypersensitivity reactions and infusion reactions etc. Incidence of Side effects of Belimumab in patients with IgG4-RD will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China